CLINICAL TRIAL: NCT06208150
Title: A Phase 3 Randomized Study Comparing Talquetamab in Combination With Pomalidomide (Tal-P), Talquetamab in Combination With Teclistamab (Tal-Tec), and Investigator's Choice of Either Elotuzumab, Pomalidomide, and Dexamethasone (EPd) or Pomalidomide, Bortezomib, and Dexamethasone (PVd) in Participants With Relapsed or Refractory Myeloma Who Have Received 1 to 4 Prior Lines of Therapy Including an Anti-CD38 Antibody and Lenalidomide
Brief Title: A Study Comparing Talquetamab Plus Pomalidomide, Talquetamab Plus Teclistamab, and Elotuzumab, Pomalidomide, and Dexamethasone or Pomalidomide, Bortezomib, and Dexamethasone in Participants With Relapsed or Refractory Myeloma Who Have Received an Anti-CD38 Antibody and Lenalidomide
Acronym: MonumenTAL-6
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64407564MMY3009; 64407564MMY3009 (Other: Janssen Research & Development, LLC); 2022-502446-27-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab; pomalidomide; elotuzumab; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Talquetamab + Pomalidomide (Tal-P) (Experimental): Participants will receive talquetamab as subcutaneous (SC) injections; pomalidomide will be self-administered as a single dose orally; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug.
  Interventions: Drug: Talquetamab; Drug: Pomalidomide; Drug: Dexamethasone
- Arm B: Talquetamab + Teclistamab (Tal-Tec) (Experimental): Participants will receive teclistamab in combination with talquetamab both as SC injection; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug.
  Interventions: Drug: Talquetamab; Drug: Teclistamab; Drug: Dexamethasone
- Arm C: Elotuzumab+ Pomalidomide+Dexamethasone (EPd) or Pomalidomide+Bortezomib+Dexamethasone (PVd) (Active Comparator): Participants will either receive elotuzumab intravenous (IV) injection in combination with pomalidomide and dexamethasone orally; or pomalidamide orally in combination with bortezomib SC injection and dexamethasone orally as per investigator choice. Dexamethasone will be administered as a pretreatment medication.
  Interventions: Drug: Pomalidomide; Drug: Elotuzumab; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered as a SC injection.
  Other Names: JNJ-64407564; Talvey
  Arms: Arm A: Talquetamab + Pomalidomide (Tal-P); Arm B: Talquetamab + Teclistamab (Tal-Tec)
Drug: Pomalidomide — Pomalidomide will be administered orally.
  Other Names: Pomalyst; Imnovid
  Arms: Arm A: Talquetamab + Pomalidomide (Tal-P); Arm C: Elotuzumab+ Pomalidomide+Dexamethasone (EPd) or Pomalidomide+Bortezomib+Dexamethasone (PVd)
Drug: Teclistamab — Teclistamab will be administered as a SC injection.
  Other Names: JNJ-64007957; Tecvayli
  Arms: Arm B: Talquetamab + Teclistamab (Tal-Tec)
Drug: Elotuzumab — Elotuzumab will be administered intravenously.
  Other Names: Empliciti
  Arms: Arm C: Elotuzumab+ Pomalidomide+Dexamethasone (EPd) or Pomalidomide+Bortezomib+Dexamethasone (PVd)
Drug: Dexamethasone — Dexamethasone will be administered either orally or intravenously.
Drug: Bortezomib — Bortezomib will be administered as a SC injection.
  Other Names: Velcade
  Arms: Arm C: Elotuzumab+ Pomalidomide+Dexamethasone (EPd) or Pomalidomide+Bortezomib+Dexamethasone (PVd)

SUMMARY:
The purpose of this study is to compare the effectiveness of either talquetamab plus pomalidomide (Tal-P) or talquetamab plus teclistamab (Tal-Tec) with elotuzumab, pomalidomide, and dexamethasone (EPd) or pomalidomide, bortezomib, and dexamethasone (PVd).

ELIGIBILITY:
Inclusion Criteria:

* Documented multiple myeloma as defined by the criteria below: (a) multiple myeloma diagnosis according to the international myeloma working group (IMWG) diagnostic criteria (b) measurable disease at screening as assessed by central laboratory, defined by any of the following: (i) serum M-protein level greater than or equal to (>=) 0.5 gram per deciliter (g/dL); or (ii) urine M-protein level >= 200 milligram (mg) per 24 hours; or (iii) light chain multiple myeloma without measurable M-protein in the serum or the urine: serum immunoglobulin (Ig) free light chain (FLC) >= 10 milligrams per deciliter (mg/dL) and abnormal serum Ig kappa lambda FLC ratio
* Relapsed or refractory disease as defined below: a) Relapsed disease is defined as an initial response to prior treatment, followed by confirmed progressive disease (PD) by IMWG criteria greater than (>) 60 days after cessation of treatment. b) Refractory disease is defined as less than (<) 25 percent (%) reduction in M-protein or confirmed PD by IMWG criteria during previous treatment or less than or equal to (<=) 60 days after cessation of treatment
* Documented evidence of PD or failure to achieve a minimal response to the last line of therapy based on investigator's determination of response by IMWG criteria on or after their last regimen
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 at screening and immediately prior to the start of administration of study treatment
* A participant must agree not to be pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of study treatment

Exclusion Criteria:

* Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients
* Stroke, transient ischemic attack, or seizure within 6 months prior to signing informed consent form (ICF)
* Major surgery or had significant traumatic injury within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment
* A maximum cumulative dose of corticosteroids of >=140 mg of prednisone or equivalent within 14-day period before the first dose of study drug
* Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain magnetic resonance imaging (MRI) and lumbar cytology are required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 3 years 5 months
  PFS is defined as the duration from the date of randomization to either progressive disease or death, whichever comes first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 years 5 months
  ORR is defined as the percentage of participants with best overall response of partial response (PR) or better according to international myeloma working group (IMWG) response criteria.
Complete Response (CR) or Better Rate | Up to 3 years 5 months
  CR or better is defined as the percentage of participants with best overall response of CR or better according to IMWG response criteria.
Very Good Partial Response (VGPR) or Better Rate | Up to 3 years 5 months
  VGPR or better is defined as the percentage of participants with best overall response of VGPR or better rate according to IMWG response criteria.
Minimal Residual Disease (MRD)-negative CR Rate | Up to 3 years 5 months
  MRD-negative CR is defined as the percentage of participants who achieve both CR or better and MRD negativity at a threshold of 10^-5 at any timepoint after the date of randomization and before disease progression or start of subsequent antimyeloma therapy (SST).
Overall Survival (OS) | Up to 3 years 5 months
  OS is defined as the time from randomization to the date of participant's death.
Progression Free Survival on Next-line Therapy (PFS2) | Up to 3 years 5 months
  PFS2 is defined as time from randomization to progression on the next line of therapy or death, whichever comes first.
Time to Next Treatment (TTNT) | Up to 3 years 5 months
  TTNT is defined as the time from randomization to the start of SST.
Serum Concentration of Talquetamab and Teclistamab | Up to 3 years 5 months
  Serum concentration of talquetamab and teclistamab will be reported.
Number of Participants with Anti-drug Antibodies (ADAs) to Talquetamab and Teclistamab | Up to 3 years 5 months
  Number of participants with ADAs to talquetamab and teclistamab will be reported.
Time to Sustained Worsening in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by Multiple Myeloma Symptom and Impact Questionnaire (MySIm-Q) | Up to 3 years 5 months
  Time to sustained worsening in symptoms, functioning and HRQoL is defined as the interval from the date of randomization to the start date of meaningful change. The MySIm-Q is a disease-specific patient-reported outcome (PRO) assessment complementary to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 item (EORTC-QLQ-C30). It includes 17 items resulting in a symptom subscale and an impact subscale.
Time to Sustained Worsening in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by EORTC-QLQ-C30 | Up to 3 years 5 months
  Time to sustained worsening in symptoms, functioning and HRQoL is defined as the interval from the date of randomization to the start date of meaningful change. EORTC-QLQ-C30 Version 3 includes 30 items that make up 5 functional scales (physical role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea or vomiting), and 5 single symptom items (dyspnea, insomnia, appetite loss, constipation, and diarrhea) and a single impact item (financial difficulties). The recall period is 7 days ("past week"), and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level.
Time to Sustained Worsening in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by EuroQol Five Dimension Questionnaire 5-Level (EQ-5D-5L) | Up to 3 years 5 months
  Time to sustained worsening in symptoms, functioning and HRQoL is defined as the interval from the date of randomization to the start date of meaningful change. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain or discomfort, and anxiety or depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time to Sustained Worsening in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by Patient Global Impression -Severity (PGI-S) | Up to 3 years 5 months
  Time to sustained worsening in symptoms, functioning and HRQoL is defined as the interval from the date of randomization to the start date of meaningful change. The PGI-S will be used as an anchor, external criterion, to determine meaningful change in scores for the MySIm-Q and EORTC-QLQ-C30 in this population. The response options are presented as a 5-point verbal rating scale from "none" to "very severe."
Time to Sustained Worsening in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by Epstein Taste Survey | Up to 3 years 5 months
  Time to sustained worsening in symptoms, functioning and HRQoL is defined as the interval from the date of randomization to the start date of meaningful change. The epstein taste survey consists of 17 items from the full 71 item PRO instrument, specific to taste changes developed for use in patients with head and neck cancer as a composite of the Vanderbilt Head and Neck Symptom Survey.
Change from Baseline in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by MySIm-Q | Up to 3 years 5 months
  Change from baseline in symptoms, functioning, and HRQoL as assessed by MySIm-Q will be reported. The MySIm-Q is a disease-specific patient-reported outcome (PRO) assessment complementary to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 item (EORTC-QLQ-C30). It includes 17 items resulting in a symptom subscale and an impact subscale.
Change from Baseline in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by EORTC-QLQ-C30 | Up to 3 years 5 months
  Change from baseline in symptoms, functioning, and HRQoL as assessed by EORTC-QLQ-C30 will be reported. The EORTC-QLQ-C30 Version 3 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea or vomiting), and 5 single symptom items (dyspnea, insomnia, appetite loss, constipation, and diarrhea) and a single impact item (financial difficulties). The recall period is 7 days ("past week"), and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high or healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale or item represents a high level of symptomatology or problems.
Change from Baseline in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by EQ-5D-5L | Up to 3 years 5 months
  Change from baseline in symptoms, functioning, and HRQoL as assessed by EQ-5D-5L will be reported. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain or discomfort, and anxiety or depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by PGI-S | Up to 3 years 5 months
  Change from baseline in symptoms, functioning, and HRQoL as assessed by PGI-S will be reported. The PGI-S will be used as an anchor, external criterion, to determine meaningful change in scores for the MySIm-Q and EORTC-QLQ-C30 in this population. The response options are presented as a 5-point verbal rating scale from "none" to "very severe."
Change from Baseline in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by Epstein Taste Survey | Up to 3 years 5 months
  Change from baseline in symptoms, functioning, and HRQoL as assessed by epstein taste survey will be reported. The epstein taste survey consists of 17 items from the full 71 item PRO instrument, specific to taste changes. developed for use in patients with head and neck cancer as a composite of the Vanderbilt Head and Neck Symptom Survey.
Percentage of Participants With Meaningful Improvement in HRQoL as Assessed by EORTC-QLQ-C30 | Up to 3 years 5 months
  Percentage of participants with meaningful improvement in HRQol as assessed by EORTC-QLQ-C30 will be reported. The EORTC-QLQ-C30 Version 3 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea or vomiting), and 5 single symptom items (dyspnea, insomnia, appetite loss, constipation, and diarrhea) and a single impact item (financial difficulties). The recall period is 7 days ("past week"), and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high or healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale or item represents a high level of symptomatology or problems.
Number of Participants with Adverse Events (AEs) by Severity | Up to 3 years 5 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. by using standard grades as follows: Grade 1: Mild; asymptomatic or mild symptoms; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; Grade 3: Severe but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening consequences; and Grade 5: Death related to AE.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (241):
- United States (48):
  - UCSF Fresno, Clovis, California
  - UCLA, Santa Monica, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Memorial Healthcare System, Hollywood, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - City of Hope Cancer Center, Newnan, Georgia
  - Kootenai Health, Coeur d'Alene, Idaho
  - University of Iowa Health Care, Waukee, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Luminis Health Center for Cancer and Blood Disorders, Annapolis, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Louis Stokes Cleveland VA Med Ctr, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - Penn State Milton S Hershey Medical Ctr, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University Of Pittsburgh Medical Center UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours Saint Francis Cancer Center, Greenville, South Carolina
  - UT Southwestern Parkland Hospital, Dallas, Texas
  - UT Southwestern, Dallas, Texas
  - Houston Methodist Neal Cancer Center at Texas Medical Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - NorthWest Medical Specialties, PLLC, Tacoma, Washington
  - Gundersen Health System, La Crosse, Wisconsin
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Fundaleu, Buenos Aires
  - Hospital Aleman, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
- Australia (7):
  - Royal Adelaide Hospital, Adelaide
  - Box Hill Hospital, Box Hill
  - St Vincents Hospital, Darlinghurst
  - St Vincents Hospital Melbourne, Fitzroy
  - Gold Coast University Hospital, Southport
  - Perth Blood Institute, West Perth
  - Wollongong Hospital, Wollongong
- Austria (3):
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Klinik Ottakring, Vienna
  - Medical University Vienna MUV, Vienna
- Belgium (4):
  - Grand Hopital De Charleroi Site Les Viviers, Charleroi
  - Ziekenhuis Oost-Limburg, Genk
  - Ghent University Hospital, Ghent
  - AZ Nikolaas - Campus Sint-Niklaas Moerland, Sint-Niklaas
- Brazil (13):
  - Cetus Oncologia, Belo Horizonte
  - DF Star, Brasília
  - Fundacao Universidade de Caxias do Sul, Caxias do Sul
  - Hospital Erasto Gaertner- Liga Paranaense de Combate ao Cancer, Curitiba
  - Hospital De Clinicas De Porto Alegre, Porto Alegre
  - Instituto D Or de Pesquisa e Ensino IDOR, Recife
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Clinica Medica Sao Germano S/S LTDA, São Paulo
  - Instituto D Or de Pesquisa e Ensino, São Paulo
- Canada (7):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - CIUSSS de l Est de l Ile de Montreal Installation Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- China (28):
  - Beijing Chaoyang Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The Second Xiangya Hospital of Central South Hospital, Changsha
  - Changzhou No 2 Peoples Hospital, Changzhou
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Fujian Meidical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Sun Yat Sen University Cancer Center, Guangzhou
  - Nanfang Hospital of Southern Medical Hospital, Guangzhou
  - First hospital affiliated of Zhejiang Medical university, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - The Affiliated Hospital of Inner Mongolia Medical College, Hohhot
  - Qilu Hospital of Shandong University, Jinan
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Ruijing Hospital Affiliated To Shanghai Jiaotong University School Of Medicine, Shanghai
  - Tongji Hospital of Tongji University, Shanghai
  - Shanghai Fourth People s Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Shanxi Bethune Hospital, Taiyuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The first affiliated hospital of xiamen university, Xiamen
- Czechia (4):
  - Fakultni nemocnice Brno, Brno-Bohunice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense C
  - Vejle Hospital, Vejle
- France (10):
  - Hopital Claude Huriez, Lille
  - CHU de Limoges Hopital Dupuytren, Limoges
  - Institut Paoli Calmettes, Marseille
  - CHU Nantes, Nantes
  - Hopital Saint Louis, Paris
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - Institut de Cancerologie Strasbourg Europe ICANS, Strasbourg
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHRU Tours Hopital Bretonneau, Tours
- Germany (7):
  - Klinikum Augsburg, Augsburg
  - Universitaetsklinikum Halle Saale, Halle
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Magdeburg A.oe.R, Magdeburg
  - Klinikum rechts der Isar der TU Muenchen, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (3):
  - 251 Airforces Hospital, Athens
  - Alexandra General Hospital of Athens, Athens
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
- Hungary (5):
  - Semmelweis Egyetem, Belgyogyaszati es Hematologiai Klinika, Budapest
  - Del Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet Szent Laszlo Telephely, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szabolcs Szatmar Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- India (3):
  - Fortis Memorial Research Institute, Gūrgaon
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
- Israel (5):
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Carmel Medical Center, Haifa
  - Rabin Medical center - Petah-Tikva, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo Alessandria, Alessandria
  - A O U Sant Orsola Malpighi, Bologna
  - oncologia medica - Oncology, Brindisi
  - ARNAS Garibaldi P O Nesima, Catania
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Asst Ovest Milanese - Ospedale Di Legnano, Legnano
  - Fondazione IRCCS Ca Granda Ospedale Policlinico Di Milano, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Presidio Ospedaliero Pescara, Pescara
  - Ospedale S. Maria Delle Croci, Ravenna
  - Oncologia Medica-Città Della Salute E Della Scienza Di Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (20):
  - Juntendo University Hospital, Bunkyō City
  - Fukuoka University Hospital, Fukuoka
  - Hamamatsu University Hospital, Hamamatsu
  - Kanazawa University Hospital, Kanazawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - National Hospital Organization Nagasaki Medical Center, Nagasaki
  - Japanese Red Cross Narita Hospital, Narita
  - Niigata Cancer Center Hospital, Niigata
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - Japanese Red Cross Osaka Hospital, Osaka
  - Sapporo City General Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Japanese Red Cross Medical Center, Shibuya-ku
  - Iwate Medical University Hospital, Shiwa-gun
  - The University of Osaka Hospital, Suita
  - Shizuoka Cancer Center, Sunto Gun
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Tottori University Hospital, Tottori
  - University of Tsukuba Hospital, Tsukuba
  - Kanagawa Cancer Center, Yokohama
- Mexico (3):
  - Centro de Quimioterapia e Investigacion, Guadalajara
  - Hematologica Alta Especialidad, Huixquilucan
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Netherlands (5):
  - Flevoziekenhuis, Almere Stad
  - Catharinaziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Haga ziekenhuis, The Hague
  - Isala Kliniek, Zwolle
- Poland (6):
  - Wojewodzki Szpital Specjalistyczny, Biała Podlaska
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Centrum Onkologii Ziemii Lubelskiej, Lublin
  - Uniwersytecki Szpital Kliniczny Nr 1 PUM im prof Tadeusza Sokolowskiego w Szczecinie, Szczecin
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Saudi Arabia (3):
  - King Abdullah International Medical Research Center (KAIMRC), Riyadh
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - King Fahad Medical City, Riyadh
- South Korea (7):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (14):
  - Hosp. de Cabuenes, Asturias
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Burgos, Burgos
  - Hosp. San Pedro de Alcantara, Cáceres
  - Hosp. Univ. Donostia, Donostia / San Sebastian
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. Univ. Lucus Augusti, Lugo
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Clinica Univ. de Navarra, Pamplona
  - Complejo Hosp de Navarra - Hosp de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
- Sweden (4):
  - Skanes universitetssjukhus, Lund
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
  - Varberg Hospital, Varberg
- Turkey (Türkiye) (5):
  - Ankara University Medical Faculty, Ankara
  - Liv Hospital Ankara, Ankara
  - Pamukkale University Medical Faculty, Denizli
  - Medipol University Hospital, Istanbul
  - Ondokuz Mayis University, Samsun
- United Kingdom (8):
  - Blackpool Victoria Hospital, Blackpool
  - University Hospital of Wales, Cardiff
  - Ninewells Hospital, Dundee
  - St James University Hospital, Leeds
  - Kings College Hospital, London
  - Nottingham City Hospital, Nottingham
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency